CLINICAL TRIAL: NCT00138788
Title: To Determine Which of Two Radiotherapy Brain Fractionation Schemes is Superior in the Treatment of Brain Metastases
Brief Title: Brain Metastases Study: Radiotherapy Fractionation Schemes in the Treatment of Brain Metastases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St George Hospital, Australia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 95/29 Graham
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2008-11-20 (Estimated); Status verified 2008-11

CONDITIONS: Neoplasm Metastasis; Brain Neoplasms
Keywords: Radiotherapy; Qualify of life; Neoplasm metastasis of the brain
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms | interventions — Chemical Fractionation

INTERVENTIONS:
Procedure: Radiotherapy, dose fractionation

SUMMARY:
This is a comparison of radiotherapy fractionation schemes for brain metastasis.

DETAILED DESCRIPTION:
Untreated brain metastases are usually fatal within a few weeks. The standard treatment for brain metastases is whole brain irradiation. This results on average in an increase in survival by 2 to 4 times compared to withholding irradiation. The majority of patients experience improvement in the level of functioning as a result of irradiation. None-the-less approximately half of patients die because of progression of the brain metastases and their quality of life is often dominated by the effects of brain metastases.

Various different dosages of radiation have been assessed and we wish to further investigate this by comparing a less intense schema with a more intense schema. Both of these fall within the range of published experience but have not been directly compared. The more intense schema may have more effect on the tumour but previous variations of dose intensity have not shown significant differences in survival. Differences in control of the metastases in the brain have been suggested but there have been no good comparisons of quality of life. Obviously when survival is measured on average in only 3 to 6 months, this is an important parameter for comparison.

Comparisons: Stratification is by diagnosis either excision or biopsy/clinical. Patients will be randomised to receive either 40Gy 20#bd or 20Gy 4#daily.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status 0 - 2.
* Brain metastasis. Brain biopsy not obligatory if known previous malignancy and multiple lesions typical on computed tomography (CT) scan of brain. Solitary lesions, if suitably located, should be biopsied and preferably excised.
* Extracranial disease stable or absent (i.e. no progression over 2 months) OR concurrent presentation of brain metastasis and extracranial disease at time of initial cancer diagnosis.
* Able to consent
* Life expectancy exceeds 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 1996-02; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Progression free survival
Quality of life

SECONDARY OUTCOMES:
Cost effectiveness
Toxicity
Neurological functioning
Survival

CONTACTS AND LOCATIONS:
Overall Officials: Associate Professor Peter H Graham, Principal Investigator — Cancer Care Centre, St George Hospital, Sydney, Australia
Locations (1):
- Cancer Care Centre, St George Hospital, Sydney, New South Wales, Australia